CLINICAL TRIAL: NCT02263469
Title: An Open Multi-centre Phase III Study to Investigate the Safety and Efficacy of Replenine®-VF in Severe Haemophilia B Patients Under the Age of 6 Years
Brief Title: A Study to Investigate the Safety and Efficacy of Replenine®-VF in Haemophilia B Patients Under the Age of 6 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: R9VF03
Record Dates: First submitted 2014-09-02; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-08

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

ARMS (1):
- Replenine®-VF (Experimental)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)

INTERVENTIONS:
Biological: Replenine®-VF (High Purity Factor IX)

SUMMARY:
The objective of this study was to assess the safety and efficacy of Replenine®-VF in children enrolled in the study, under the age of six years, with severe haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Patients under six years of age at the time of entry with severe Haemophilia B at the time of diagnosis without inhibitors to FIX and requiring Factor IX therapy.

Exclusion Criteria:

-

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-08; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Amount of Factor IX Administered per Month (IU/KG) | 26 Weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Oddzial Pediatrii, Hematologii I Onkologii, ul. Marszalkowska 24, 00-576, Warsaw, Poland
- Ukraine (3):
  - Institute of Urgent and Recovery Surgery, Academy of Medical Science of Ukraine, Leninski Avenue, Donetsk
  - Institute of Haematology and Transfusiology, Academy of Medical Science of Ukrainem Berlynskogo Str., Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Academy of Medical Science of Ukraine, Gen. Chuprynkea Str., Lviv

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk